CLINICAL TRIAL: NCT04692168
Title: Influence of Chemotherapy on Postural Control and Quality of Life in Women With Gynaecological Cancer: a Prospective Observational Study
Brief Title: Influence of Chemotherapy on Postural Control in Women With Cancer
Status: Completed | Type: Observational
Sponsor: Aline Reinmann (Other)
Responsible Party: Sponsor-Investigator, Aline Reinmann, Principal Investigator, School of Health Sciences Geneva
Organization: School of Health Sciences Geneva (Other)
Other Study IDs: 105909; 2020-01639 (Registry Identifier: BASEC)
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Cancer, Breast; Cancer, Gynecologic
Keywords: postural control; balance; chemotherapy induced peripheral neuropathy; quality of life
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Entire group: The group will be test prior and three months after a neurotoxic chemotherapy for gynecological cancer.

SUMMARY:
The aim of this study is to understand the strategies for adapting postural control in patients who have received chemotherapy treatment for gynaecological cancer.

DETAILED DESCRIPTION:
Chemotherapy can cause many side effects, including peripheral neuropathies. Chemotherapy induced peripheral neuropathies (CIPN) are primarily sensory impairments that can alter the signals for somatosensory feedback and thus affect the postural control in the standing position. The objective of this study is to evaluate the impact of chemotherapy and peripheral neuropathies on postural control in the standing position. As balance maintenance is a complex construct involving different systems, this study will evaluate maintenance strategies during sensory disturbances in order to better understand post-chemotherapy coping strategies. These sensory disturbances concern vision (eyes closed) and the alteration of the somatosensory system (foam under the feet and vibration system). In addition, this study will evaluate balance in double task situations and dynamic stability. Given the consequent impact of chemotherapy and peripheral neuropathies on quality of life, a quality of life questionnaire will also be administered.

ELIGIBILITY:
Inclusion Criteria:

Women

* between 18 and 65 years;
* with a gynaecological cancer about to start chemotherapy known to be neurotoxic (paclitaxel, docetaxel, nab-paclitaxel, or paclitaxel-carboplatin);
* able to stand upright for 30 s on a flat surface without assistance;
* able to provide written consent

Exclusion Criteria:

Women

* with pre-existing vestibular, uncorrectable visual, or somatosensory disorders or other pathologies altering postural control that would influence testing;
* with exposure to known neurotoxic chemotherapy (paclitaxel, docetaxel, nab-paclitaxel, vinorelbine, trastuzumab-emtansine, eribulin, or paclitaxel-carboplatin) that may have caused previous CIPN;
* with an inability to perform the test due to poor comprehension of instructions or psychological problems.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 31 women between the ages of 18 and 65 consulting at the University Hospitals for their oncological disease.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline : postural control under various conditions. | Prior and three months after chemotherapy
  The postural control will be assessed by a force platform. Three 30-second tests will be performed for each test condition. The test conditions are as follows: eyes open, eyes closed, firm surface, soft surface, with vibrator, without vibrator, with dual task. The test position will be standing with the feet 10 cm apart at heel level and 15 cm apart at hallux level, with the arms along the body, fixing a point on the wall at 0.90 cm. Parameters of center of pressure and strength will be recorded at a frequency of 100 Hertz.

SECONDARY OUTCOMES:
Change from baseline : modifications of postural control according to the conditions tested. | Prior and three months after chemotherapy
  The postural control will be assessed by a force platform. Three 30-second tests will be performed for each test condition. The test conditions are as follows: eyes open, eyes closed, firm surface, soft surface, with vibrator, without vibrator, with dual task. The test position will be standing with the feet 10 cm apart at heel level and 15 cm apart at hallux level, with the arms along the body, fixing a point on the wall at 0.90 cm. Parameters of center of pressure and strength will be recorded at a frequency of 100 Hertz.
Change from baseline : standing dynamic stability. | Prior and three months after chemotherapy
  The standing dynamic stability will be assessed by a force platform with the limits of stability test (LOS). The test position will be standing with the feet 10 cm apart at heel level and 15 cm apart at hallux level, with the arms along the body, fixing a computer at a distance of 0.90 cm. Parameters of center of pressure and strength will be recorded at a frequency of 100 Hertz.
Change from baseline : quality of life assessed by the questionnaire Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-NTX). | Prior and three months after chemotherapy
  The FACT/GOG-NTX was chosen to assess the quality of life (QoL). This questionnaire assesses physical well-being, family/social well-being, emotional well-being, functional well-being and other concern. Participants will have to answer the different statements by ticking the box corresponding to what they feel is adequate between 0 (not at all) and 4 (a lot). The minimum score is 0 and the maximum score is 152. The higher the score, the better the QoL.
Change from baseline : investigate the association between the severity of CIPN (mild, moderate, severe) and the postural control, dynamic balance and QoL of individuals with gynaecological cancer. | Prior and three months after chemotherapy
  The clinical version of the Total Neuropathy Score will be used to evaluate the presence of peripheral neuropathy. A test of superficial sensitivity, vibration sensitivity, reflexes and strength will be carried out. The minimum score is 0 and the maximum score is 24. A score between 0 and 8 indicates mild peripheral neuropathy, between 9 and 16 a moderate peripheral neuropathy and above 17 a severe neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Reinmann, Principal Investigator — School of Health Sciences Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes will be made available.
Time Frame: Data will be available within 6 months of study completion
Access Criteria: At the end of the project the data will be deposited in the Yareta repository developed by the University of Geneva OR in an institutional repository. This choice will ensure that data is archived and shared in accordance with FAIR principles (Findability, Accessibility, Interoperability, and Reuse of digital assets).

REFERENCES:
- [Background] Kneis S, Wehrle A, Freyler K, Lehmann K, Rudolphi B, Hildenbrand B, Bartsch HH, Bertz H, Gollhofer A, Ritzmann R. Balance impairments and neuromuscular changes in breast cancer patients with chemotherapy-induced peripheral neuropathy. Clin Neurophysiol. 2016 Feb;127(2):1481-1490. doi: 10.1016/j.clinph.2015.07.022. Epub 2015 Aug 14. PMID 26350407
- [Background] McCrary JM, Goldstein D, Trinh T, Timmins HC, Li T, Menant J, Friedlander M, Lewis CR, Hertzberg M, O'Neill S, King T, Bosco A, Harrison M, Park SB. Balance Deficits and Functional Disability in Cancer Survivors Exposed to Neurotoxic Cancer Treatments. J Natl Compr Canc Netw. 2019 Aug 1;17(8):949-955. doi: 10.6004/jnccn.2019.7290. PMID 31390588
- [Background] Monfort SM, Pan X, Loprinzi CL, Lustberg MB, Chaudhari AMW. Impaired Postural Control and Altered Sensory Organization During Quiet Stance Following Neurotoxic Chemotherapy: A Preliminary Study. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419828823. doi: 10.1177/1534735419828823. PMID 30741022
- [Background] Muller J, Ringhof S, Vollmer M, Jager LB, Stein T, Weiler M, Wiskemann J. Out of balance - Postural control in cancer patients before and after neurotoxic chemotherapy. Gait Posture. 2020 Mar;77:156-163. doi: 10.1016/j.gaitpost.2020.01.012. Epub 2020 Jan 15. PMID 32036320
- [Derived] Reinmann A, Bodmer A, Koessler T, Gligorov J, Bruyneel AV. Postural control impairments following neurotoxic chemotherapy in women with cancer: a prospective observational study. BMC Womens Health. 2025 May 30;25(1):269. doi: 10.1186/s12905-025-03790-4. PMID 40448057
- [Derived] Reinmann A, Bruyneel AV, Gligorov J, Mesure S, Combescure C, Koessler T, Bodmer A. Influence of chemotherapy on postural control and quality of life in women with gynaecological cancer: a protocol of a prospective observational study. BMJ Open. 2022 Sep 7;12(9):e061664. doi: 10.1136/bmjopen-2022-061664. PMID 36691184